CLINICAL TRIAL: NCT04381884
Title: A Pilot, Proof of Concept Trial to Prove Ivermectin Efficacy in the Reduction of SARS-CoV-2 Replication at Early Stages of COVID-19
Brief Title: Ivermectin Effect on SARS-CoV-2 Replication in Patients With COVID-19
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Laboratorio Elea Phoenix S.A. (Industry)
Collaborators: Universidad Nacional de Salta (Other); Centro de Investigación Veterinaria Tandil CIVETAN (Unknown); Fundación Hospital de Pediatría Prof. Dr. Juan P. Garrahan (Other); Universidad Nacional de Quilmes (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IVM-AR-1
Record Dates: First submitted 2020-05-05; First posted 2020-05-11 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-10

CONDITIONS: COVID-19 Drug Treatment
Keywords: COVID-19; IVERMECTIN; SARS-CoV-2 viral load
MeSH Terms: conditions — COVID-19 | interventions — Ivermectin

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to receive Ivermectin 600 µg / kg / once daily plus standard care or standard care upon diagnosis of COVID-19.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- IVERMECTIN (IVER P®) (Experimental): Patients in this group will receive Ivermectin (IVER P®) 600 µg / kg / once daily plus standard care.
  Interventions: Drug: IVERMECTIN (IVER P®) arm will receive IVM 600 µg / kg once daily plus standard care. CONTROL arm will receive standard care.
- CONTROL (No Intervention): Patients in this group will receive standard care.

INTERVENTIONS:
Drug: IVERMECTIN (IVER P®) arm will receive IVM 600 µg / kg once daily plus standard care. CONTROL arm will receive standard care. — IVERMECTIN (IVER P®) arm will receive IVM 600 µg / kg once daily plus standard care. CONTROL arm will receive standard care.
  Arms: IVERMECTIN (IVER P®)

SUMMARY:
In the context of COVID-19 pandemic, a report on ivermectin suppression of SARS-CoV-2 viral replication in cell cultures has been published, and the use of this medication seems to be potentially useful for the therapy. IVM safety profile and IVM wide spectrum enables to move forward with the investigation in patients infected by SARS-CoV-2 as a proof-of-concept of its possible use in the management of patients with COVID-19, given the current pandemic situation.

DETAILED DESCRIPTION:
Ivermectin (IVM) is a semisynthetic antiparasitic agent belonging to the avermectin group, drugs isolated from Streptomyces avermitilis. Ivermectin is widely used for humans and animals, with millions of doses annually administered through mass drug distribution programs held by the World Health Organization (WHO - 2016). Since 1980, Ivermectin has been included in the Essential Medicines List of the World Health Organization (WHO - 2019).

This medicine is orally administered and is usually used for the treatment against nematodes and ectoparasites, making this drug the first-choice medication for onchocerciasis, lymph filariasis, itch and strongylosis.

Until now, SARS-CoV-2 viral load dynamics has not been clearly determined. However, works tending to a preliminary characterization of the viral load (VL) behavior have emerged. One of them, the most substantial one, includes the work done by Kai-Wang showing the VL behavior during the 30 days before the onset of COVID-19 symptoms (Kai-Wang To et al; 2020). In this work, an average of 7.5 oropharyngeal samples of individuals with severe (n=10) and moderate (n=13) COVID-19 have been assessed. Time between the onset of symptoms and hospitalization ranged between 0 and 13 days, with a mean of 4 days. VL median at day 0 in all patients was 5.2 log10 copies/mL, and no significant differences between severe and moderate COVID-19 groups occurred. The viral load peak observed during the first week from the onset of symptoms had a median equal to 6.91 (Q1-Q3: 4.27-7.40) and 5.29 (Q1-Q3: 3.91-7.56) log10 copies/mL in severe and moderate COVID-19 patients, respectively. There was no significant difference between both groups (p=0.52). Likewise, no difference between patients with and without comorbidities has been observed (n of patients equal to 12 and 11, respectively) as per initial VL (p=0.49) and peak VL (p=0.29). However, it has been observed that the VL peak was directly associated with the age of the patient (R2=0.48 and p=0.02). In a combined analysis of all patients (n=23), it has been observed that the VL grows in the first days following the onset of symptoms and that, in the 5-6 days, VL falls sharply, reaching a lower mean value, yet similar to that of the day 0. General VL behavior from day 9 to 30 showed a negative slope (VL fall) equal to -0.15 (95% confidence interval: -0.19 to -0.11) log10 per daya. It must be emphasized that by day 20 from the onset of symptoms, VL mean continues to be quantifiable (4 log10 copies/mL), and that 7/23 (30%) patients show viral RNA detection after such day.

In other paper, the VL of 17 patients with an age median of 59 (range 26-76 years) has been studied, who tested positive for SARS-CoV-2 (Zou et al; 2020). Nonetheless, VL measurement by nasal swab was performed in 16 patients and quantification was conducted relatively, expressed in Ct values (cycle threshold), which is related with the VL copies detected in the molecular reaction: the lower the Ct value, the greater the VL, and vice versa. The feature worth noting of such work is that VL dynamics varies widely from one patient to another. Contrary to the work of Kai-Wang To et al. [1], the VL peak seems to occur earlier (first three days), whereas the sharp VL fall is at day 6 approximately, from which day the VL is undetectable in most patients. Only very few patients show detectable viral RNA after 10 days from the onset of symptoms.

In other work, pharyngeal swabs performed in 67 patients have been studied (Pan et al; 2020). VL dynamics similar to that reported by Kai-Wang To et al. is observed, with a VL of approximately 4 to 5 log10 copies/mL at day 0 of the onset of symptoms, a peak at day 6/7 (8 log10 copies/mL) and a sharp fall from day 8 of the onset of symptoms. A temporary onset of viremia is observed with a VL of 4 log10 copies/mL up to day 15 from the onset of symptoms.

Finally, in the work published by Wölfel et al. [4] much more accelerated dynamics than that in the work of Kai-Wang To et al. and Pan et al. (Wölfel et al; 2020) is observed, and the peak appearing much earlier than the day 4 from the onset of symptoms in the nine studied patients. Additionally, in 8 patients, the VL falls sharply reaching values below the quantification limit (2 log10 copies/mL) at day 10-11 following the onset of symptoms. Although there are transient VL relapses after day 10, this value remains very close to the study quantification limit.

In conclusion, if the works of Kai-Wang and Pan are considered, a greater viral RNA half-life is expected at day 10 following the onset of symptoms. Even though in the works of Zou and Wölfel the peak occurs much earlier than the first five days and viral negativity occurs after day 10-11 following the onset of symptoms. Method variability among the many works is a limiting factor when comparing the outcomes. That is why, due to the sample size in Kai Wang et al (n=23) and Zou et al (n=67), it is suggested to use these works as reference and to consider the works of Pan (n=17) and Wölfel (n=9) as part of behavior diversity. It is important to define the period in which therapy is to be initiated from the onset of symptoms so that the sharp fall observed post-peak is not a factor that biases the potential antiviral effect of the drug.

Considering these backgrounds along with the preliminary study with ivermectin, it is not possible to define a specific, progressive outcome for the reduction of the VL, but it may be expressed in a variation percentage with respect to the control population (without therapy) at the end of treatment. This percentage difference between the treated population and the untreated population must be greater than the variation observed for the study day or period in the patients included in the above mentioned works, since such percentage difference would replicate the behavior in our control population.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of both genders, aged between 18 and 69.
2. Patients infected by SARS-CoV-2 confirmed by PCR.
3. Hospitalized patients with symptoms onset 5 days before executing the Informed Consent.
4. No comorbidities affecting the patient´s prognosis, rendering them high risk patients.
5. Documented acceptance to participate by means of the execution of the Informed Consent.
6. Female patients of childbearing age must have a negative pregnancy test and must use adequate contraceptive methods (for example, intrauterine devices, hormonal contraceptives, barrier methods, chastity or tubal ligation) during their participation in the study and for one month after the last medication dose in the case of those receiving ivermectin.

Exclusion Criteria:

1. Allergy or hypersensitivity to ivermectin and/or its inactive ingredients.
2. Patients meeting COVID-19 severity criteria, with respiratory distress or requiring intensive care.
3. Using medications having potential activity against SARS-CoV-2 such as hydroxychloroquine, chloroquine, lopinavir, ritonavir, remdesivir, azithromycin in the last 3 months.
4. Use of immunodepressants (including systemic corticosteroids) in the last 30 days.
5. Known HIV infection with CD4 count <300 cell/µL.
6. Pregnant or lactating patients.
7. Patients with other acute infectious diseases.
8. Patients with medical conditions such as malabsorption syndromes affecting proper ivermectin absorption.
9. Patients with acute allergy conditions or with severe allergic reactions background.
10. Patients with autoimmune disease and/or decompensated chronic diseases.
11. Patients with uncontrolled, intercurrent diseases including renal impairment, hepatic impairment, symptomatic congestive heart failure, unstable chest angina, heart arrhythmia or psychiatric conditions that may limit adherence to CT requirements.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2020-05-18 (Actual); Primary Completion 2020-09-29 (Actual); Study Completion 2020-09-29 (Actual)

PRIMARY OUTCOMES:
Reduction in SARS-CoV-2 viral load | 1 - 5 days
  Number of patients in whom the SARS-CoV-2 viral load decreases after Ivermectin treatment

SECONDARY OUTCOMES:
Number of patients with partial or complete response in COVID-19 clinical symptoms | 1 - 7 days
  Clinical symptoms will be assessed after the treatment with the study drug
Number of patients with worsening in the clinical condition | 1 - 7 days
  Effect of Ivermectin therapy on severity indicators such as need of intensive care unit and assisted ventilation, or mortality
Number of patients with adverse events as a measure of safety and tolerability | 1 month
  Ivermectin safety profile will be evaluated according to Common Terminology Criteria for Adverse Events (CTCAE version 4.0)
Ivermectin concentrations measured in plasma | 1 month
Evaluation of reactivity of the antibodies against SARS-CoV-2 | 1 month
  Effect of Ivermectin therapy on the onset of SARS-CoV-2 antibodies through the determination of serological changes

OTHER OUTCOMES:
Observed effects to Ivermectin serum concentrations quantified at different treatment time points. | 1 month

CONTACTS AND LOCATIONS:
Locations (3):
- Argentina (3):
  - Hospital de Cuenca Alta, Cañuelas, Buenos Aires
  - Centro de Educación Médica e Investigaciones Clínicas "Norberto Quirno" CEMIC, Buenos Aires, Buenos Aires F.D.
  - Hospital de Infecciosas Francisco Javier Muñiz, Buenos Aires

REFERENCES:
- [Derived] Krolewiecki A, Lifschitz A, Moragas M, Travacio M, Valentini R, Alonso DF, Solari R, Tinelli MA, Cimino RO, Alvarez L, Fleitas PE, Ceballos L, Golemba M, Fernandez F, Fernandez de Oliveira D, Astudillo G, Baeck I, Farina J, Cardama GA, Mangano A, Spitzer E, Gold S, Lanusse C. Antiviral effect of high-dose ivermectin in adults with COVID-19: A proof-of-concept randomized trial. EClinicalMedicine. 2021 Jun 18;37:100959. doi: 10.1016/j.eclinm.2021.100959. eCollection 2021 Jul. PMID 34189446